CLINICAL TRIAL: NCT02839967
Title: Influence of Intraoral Photobiomodulation on Pain, Joint Mobility, Functionality and Quality of Life in Individuals With Temporomandibular Joint Dysfunction
Brief Title: Influence of Intraoral Photobiomodulation in Individuals With Temporomandibular Joint Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Daniela Ap. Biasotto-Gonzalez, Doctor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PHOTOBIOMODULATION DTM INT.
Record Dates: First submitted 2015-09-29; First posted 2016-07-21 (Estimated); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Temporomandibular Disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Photobiomodulation group (Experimental): For the purposes of photobiomodulation is used a portable cluster 9 PainAway ® diodes manufactured by Multi Radiance Medical ® (Solon, OH-USA), and 1 905 nm diode LASER, 4 875 nm LED diodes and 4 670 nm diodes LED, 4 cm2 beam, emitting an energy of 39.27 J.
  Interventions: Other: Photobiomodulation
- Photobiomodulation placebo group (Placebo Comparator): To provide the "blinding" of the participants of the study we will use two identical photobiomodulation equipment supplied by the manufacturer, being an active and another a placebo, but both have identical light and sound device (do not send energy and heat, non-coherent light without biological effect). The devices are named in X and Y for a researcher who does not participate in treatment and assessments.
  Interventions: Other: Photobiomodulation placebo

INTERVENTIONS:
Other: Photobiomodulation — Intraoral photobiomodulation is applied in the temporal, medial and lateral pterygoid, bilateral, totaling 4 points of application of phototherapy. The researcher who will perform the treatments will receive the equipment with the stylus activates and pre-programmed dose, an eye protection (glasses, opaque) will be used by the participants, to protect the eyes, because the same does not cause any sensation to volunteer. The technique is used, contact an area. The individual is positioned supine on a stretcher, with the legs supported on a foam roller 20 cm in diameter, the head supported on a pillow, to accommodate her comfortably in a resting posture, prompted the opening of the mouth and placing the tip of photobiomodulation in sections as described below, with 2 minutes interval between one application and another for rest with the mouth closed.
  Arms: Photobiomodulation group
Other: Photobiomodulation placebo — The volunteers will be subjected to the same Group intervention, Photobiomodulation and the researcher will receive the equipment unaware if the pen that will apply the phototherapy is active or placebo, only the research coordinator will have this knowledge, and for this group the researcher will receive placebo pen. Fits the caveat that, when the voluntary participation, will be held with the active pen treatment.
  Arms: Photobiomodulation placebo group

SUMMARY:
According to the International Association for the Study of Pain (IASP), the temporomandibular pain and dysfunction syndrome (TMD) is characterized as a subset of orofacial pain, whose signs and symptoms include pain or discomfort in the temporomandibular joints. Pain is considered one of the most common and limiting clinical manifestations. One of the most used resources to treat muscle pain is the low-level laser therapy (LLLT), However, the mechanisms responsible for the effects observed in clinical trials remain poorly elucidated, as well as therapy with light emitting diode therapy (LEDT) which, has some advantages, among them the larger area radiation point and low cost. However, its effects remain elusive in intraoral application in temporal muscle, lateral and medial pterygoid muscle. Assuming that there is need to investigate therapeutic resources that combine not only different wavelengths as well as different light sources (LED and LLLT), this study aims to evaluate the effect of photobiomodulation with a combination of different light sources on pain, joint mobility, equity and quality of jaw movements after treatment in patients with TMD. It will be made a randomized, placebo-controlled and double-blind clinical trial. Individuals participate with myogenic temporomandibular disorder, being allocated into 2 groups randomly and stratified by the method of sealed envelopes. The results will be evaluated using: RDC/TMD, digital caliper, visual analog scale, and kinematics. The protocols will be used in a 6 sessions and will be evaluated in four different moments. The analyses of the data will be performed by adopting a significance level of 5%.

ELIGIBILITY:
Inclusion Criteria:

* Women with disfunction temporomandibular.
* Limitation of mandibular opening below 40 mm.
* score of masticatory muscle pain greater than 3 cm in accordance with EVA.

Exclusion Criteria:

* women who have dental failures, total or partial prosthesis.
* systemic diseases .
* history of trauma to the face and or ATMor the ATM dislocation history.
* orthodontic treatment and/or medicated that affects the musculoskeletal system.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-09-25 (Actual); Primary Completion 2017-05-10 (Actual); Study Completion 2018-01-20 (Actual)

PRIMARY OUTCOMES:
Intensity of pain as measured by Visual analogue scale | five minutes
  Visual analogue scale is a tool which allows easy measurement of the intensity of the pain, and consists of a straight line of 10 cm in length, the ends have a verbal description (without pain and worst pain ever felt, respectively), in which the volunteers will be directed to make a perpendicular dash between the two extremes that represents the level of pain she presented at that time.
Measured by joint mobility | ten minutes
  Will be used a digital meter to assess the breadth of mandibular movement (in mm), i.e. will be measured the opening of the mouth, sides (right and left) and protrusion.

SECONDARY OUTCOMES:
Functional as measured by Patient specific Functional scale | ten minutes
  Patient specific Functional scale is a global scale, so it can be used for any region of the body. The patient is asked to identify up to 3 activities that are unable to perform or presents any difficulty and may incorporate issues that were not addressed in a generic scale but it's important for the patient's problem. The measurement is made by Likert-type scales of 11 points for each activity, and the higher the average score (0-10) the better the patient's ability to perform the activities.
quality of life measured by questionnaire (WHOQOL-BREF) | ten minutes

CONTACTS AND LOCATIONS:
Overall Officials: Daniela ap Biasotto-Gonzalez, Phd, Principal Investigator — University of Nove de Julho
Locations (1):
- University of Nove de Julho, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Herpich CM, Leal-Junior ECP, Politti F, de Paula Gomes CAF, Dos Santos Gloria IP, de Souza Amaral MFR, Herpich G, de Azevedo LMA, de Oliveira Gonzalez T, Biasotto-Gonzalez DA. Intraoral photobiomodulation diminishes pain and improves functioning in women with temporomandibular disorder: a randomized, sham-controlled, double-blind clinical trial : Intraoral photobiomodulation diminishes pain in women with temporomandibular disorder. Lasers Med Sci. 2020 Mar;35(2):439-445. doi: 10.1007/s10103-019-02841-1. Epub 2019 Jul 19. PMID 31325122